CLINICAL TRIAL: NCT06993623
Title: Heparin Binding Protein Versus Platelet Count and Mean Platelet Volume Kinetics as Indicators for Diagnosis and Prognosis of Ventilator Associated Pneumonia
Brief Title: Heparin Binding Protein Versus Platelet Count and Mean Platelet Volume Kinetics in the Diagnosis and Prognosis of VAP
Status: Not yet recruiting | Type: Observational
Sponsor: Esraa Hamdy Thabit Riad (Other)
Responsible Party: Sponsor-Investigator, Esraa Hamdy Thabit Riad, Assistant lecturer of anesthesiology and ICU, Minia University
Organization: Minia University (Other)
Other Study IDs: 1489/03/2025
Record Dates: First submitted 2025-05-01; First posted 2025-05-29 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-03

CONDITIONS: Ventilator Associated Pneumonia (VAP)
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Diagnostic Test: heparin binding protien — compare between Heparin binding protien and platelet count and mean platelet volume kinetics in diagnosis and prognosis of VAP

SUMMARY:
mechanically ventilated for 48 hours or more and subsequently develop ventilator-associated pneumonia (VAP). After obtaining approval from the local ethical committee at the Faculty of Medicine, El-Minia University, and informed consent from first-degree relatives, patients will be enrolled and classified into two groups based on clinical outcomes: Group A (survivors with successful extubation) and Group B (non-survivors with prolonged mechanical ventilation and/or 30-day mortality). Prolonged mechanical ventilation (PMV) is defined as ≥21 days of ventilation. Blood samples will be collected from participants to measure heparin-binding protein (HBP), mean platelet volume (MPV), and the MPV-to-platelet count (PC) ratio. Laboratory analysis will be blinded to the clinical outcome group to ensure objectivity. The study aims to investigate the potential of these biomarkers in predicting prognosis and guiding clinical decisions in patients with VAP.

DETAILED DESCRIPTION:
This prospective, single-blinded observational study aims to investigate the prognostic value of heparin-binding protein (HBP), mean platelet volume (MPV) kinetics, and the MPV-to-platelet count (PC) ratio in adult patients with ventilator-associated pneumonia (VAP). The study will be conducted on 80 adult patients (aged >18 and <70 years) admitted to the intensive care unit (ICU) at El-Minia University Hospitals. Eligible patients must have been mechanically ventilated for more than 48 hours and meet the diagnostic criteria for VAP based on clinical and radiological data, including a Modified Clinical Pulmonary Infection Score (CPIS) >6. The CPIS will be calculated without including microbiological culture results.

After obtaining ethical approval and informed consent from first-degree relatives, patients will be enrolled and classified retrospectively into two groups based on clinical outcomes:

Group A: Survivors (patients who undergo successful extubation).

Group B: Non-survivors (patients requiring prolonged mechanical ventilation-defined as ≥21 days-and/or those who die within 30 days of diagnosis).

Blood samples will be collected and tested for HBP, MPV kinetics, and the MPV/PC ratio. All laboratory analyses will be performed in a blinded manner to eliminate bias, as the clinical pathologist will not be informed of the patient group classification.

The primary objective of this study is to evaluate whether these biomarkers can predict clinical outcomes and assist in the risk stratification of patients with VAP.

Exclusion criteria include patients with:

Pre-existing infections or sepsis at the time of ICU admission.

Underlying conditions that may affect platelet function or morphology (e.g., cancer, chronic liver disease, end-stage renal disease).

Primary hematologic disorders, including disseminated intravascular coagulation.

Severe thrombocytopenia (platelet count ≤20×10⁹/L) or those receiving platelet transfusions.

The study aims to generate insights that may guide future prognostic and therapeutic strategies in managing critically ill patients with VAP.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients < 18 years old<70years 2. MV for more than 48 h. 3 . Signs of VAP according to clinical and radiological data , Modified Clinical Pulmonary Infection Score (CPIS) will be calculated for the patients and will be included when CPIS > 6 . Modified CPIS will be calculated without considering culture results.(12)

Exclusion Criteria:

- . Patients with pre-existing infections or sepsis at ICU admission. 2. Patients with underlying conditions such cancer, chronic liver illnesses, end-stage renal disease, etc. that may impact platelet function or morphology.

3. primary hematological disorders, disseminated intravascular coagulation. 4.severe thrombocytopenia (platelet count ≤ 20x109 L-1) and receiving platelet transfusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged 18-70 years) admitted to the intensive care unit (ICU) at El-Minia University Hospitals, who are mechanically ventilated for more than 48 hours and subsequently develop ventilator-associated pneumonia (VAP). All participants must fulfill the clinical and radiological criteria for VAP with a Modified Clinical Pulmonary Infection Score (CPIS) >6.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
HBP levels in survivors and non survivors patients of VAP measured by ng\ ml using ElISAImmunoassay | within 30 days after VAP diagnosis
  To determine whether elevated HBP levels , change in platelet count and mean platelet volume kinetics are associated with mortality and prolonged mechanical ventilation in patients with VAP.

CONTACTS AND LOCATIONS:
Locations (1):
- Minia university Hospitals, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided